CLINICAL TRIAL: NCT01610674
Title: Perioperative Diabetes Care: Developing and Testing an Implementation Strategy in Terms of Effectiveness, Experiences and Costs
Brief Title: Developing and Testing an Implementation Strategy to Improve Perioperative Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Marlies Hulscher, M.E.J.L. Hulscher, PhD, Radboud University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Diabetesperiop2008
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus; Surgery
Keywords: Diabetes mellitus; Surgery; Implementation; Quality of care; Quality indicators
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tailored improvement strategy (Experimental): In 3 hospitals a tailored strategy to improve perioperative diabetes care is performed
  Interventions: Other: Tailored improvement strategy
- Usual perioperative diabetes care (No Intervention): Three hospitals that provide usual perioperative diabetes care serve as control hospitals

INTERVENTIONS:
Other: Tailored improvement strategy — A step-wise implementation model is applied:
  1) recommendations on optimal perioperative diabetes care (e.g. the administration of intravenous insulin, encouragement of diabetes self-management) are systematically translated into quality indicators; 2a) using these quality indicators, current care is measured by performing a medical record search among 400 patients in 6 hospitals; 2b) barriers and facilitators for optimal care are measured by performing interviews with professionals 3) based on this information an implementation strategy is developed; 4) implementation activities are enacted in 3 hospitals and 5) evaluated in a controlled before-after design in 6 hospitals providing before and after intervention 400 patients.
  Arms: Tailored improvement strategy

SUMMARY:
Optimising glycaemic control during hospital stay reduces the rate of infections, length of stay and mortality, in particular in surgical patients. In this study, we test a strategy to implement optimal perioperative diabetes care in a controlled before and after design in 6 Dutch hospitals.

DETAILED DESCRIPTION:
OBJECTIVE/RESEARCH QUESTION Optimising glycaemic control during hospital stay reduces rate of infections, length of stay and mortality,in particular in surgical patients. In guidelines and literature recommendations on optimal perioperative diabetes care are described. Nevertheless, in daily practice, perioperative glycaemic control is very often not achieved. This study aims at developing an implementation strategy that is tested on feasibility to improve perioperative diabetes care in terms of effectiveness, experiences and costs.

DESIGN/OUTCOME MEASURES/IMPLEMENTATION STRATEGY A step-wise implementation model is applied: 1) recommendations on optimal perioperative diabetes care (e.g. the administration of intravenous insulin, encouragement of diabetes self-management) are systematically translated into quality indicators; 2a) using these quality indicators, current care is measured by performing a medical record search among 400 patients in 6 hospitals; 2b) barriers and facilitators for optimal care are measured by performing interviews with professionals and, e.g. regarding self-management, with patients; 3) based on this information an implementation strategy is developed;4) implementation activities are enacted and 5) evaluated in a controlled before-after design in 6 hospitals providing before and after intervention 400 patients.

DATA ANALYSIS To obtain an indication of the effectiveness of the strategy, baseline and post intervention outcomes of intervention hospitals are compared with outcomes in control hospitals, using the quality indicators. Experiences of participants in the intervention hospitals will be measured to, if necessary, adapt the strategy to make it more effective and acceptable.

ECONOMIC EVALUATION A cost analysis of the implementation strategy will take place. Implementation costs will be related to the difference in percentage of patients treated as described in the quality indicators before and after implementation. Information on the costs and effects at the patient level will also be compared before and after the implementation of the recommendations on optimal care.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus AND
* Cardiac surgery OR
* Abdominal surgery OR
* Large joint orthopedic surgery And
* Duration of surgery minimum one hour

Exclusion Criteria:

* Rejection to participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 811 (Actual)
Dates: Start 2009-01; Primary Completion 2014-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Current care study | 1 year
  the primary outcome measure is the adherence to the quality indicators (derived from international guidelines and scientific literature)
  Baseline measurement
Feasibility study | 1 year
  the primary outcome measure regarding effectiveness is the adherence to developed quality indicators
  baseline measurement and follow up measurement following improvement intervention
Barrier analysis | 1 year
  the primary outcomes in the barrier analysis are the barriers and facilitators among professionals regarding adherence to the quality indicators
  interview study

SECONDARY OUTCOMES:
current care study | 1 year
  the secondary outcome measure is the outcome of care (e.g. glycemic control) before intervention data
feasibility study | 1 year
  the secondary outcome measure is the outcome of care (e.g. glycemic control) before and after data
  the secondary outcome measures are the experiences of professionals and patients with different elements of the implementation strategy and the changed care, and the cost of the tested strategy

CONTACTS AND LOCATIONS:
Overall Officials: Marlies Hulscher, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Netherlands

REFERENCES:
- [Derived] Hommel I, van Gurp PJ, Tack CJ, Wollersheim H, Hulscher ME. Perioperative diabetes care: development and validation of quality indicators throughout the entire hospital care pathway. BMJ Qual Saf. 2016 Jul;25(7):525-34. doi: 10.1136/bmjqs-2015-004112. Epub 2015 Sep 17. PMID 26384710